CLINICAL TRIAL: NCT02831998
Title: Clinical Evaluation of the Antimicrobial Effectiveness of Topically Applied ZP
Brief Title: In-vivo Efficacy of Patient Preoperative Prep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZX-ZP-0073 / 865-105
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-06

CONDITIONS: Surgical Skin Preparation
MeSH Terms: interventions — citrate, isopropyl alcohol, methylene blue, parabens drug combination; Ethanol; Chromogranins; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZP (70% IPA) (Experimental): Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ZuraPrep
- ChloraPrep (Active Comparator): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ChloraPrep
- ZP Vehicle (Placebo Comparator): ZP without IPA
  Interventions: Drug: ZP Vehicle

INTERVENTIONS:
Drug: ZuraPrep — Apply topically.
  Other Names: Isopropyl alcohol 70%; ZP
  Arms: ZP (70% IPA)
Drug: ChloraPrep — Apply topically.
  Other Names: CHG 2%/IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: ChloraPrep
Drug: ZP Vehicle — Apply topically.
  Other Names: ZP without IPA
  Arms: ZP Vehicle

SUMMARY:
The objective of the study is to demonstrate the antimicrobial efficacy of the ZP Preoperative Prep on skin flora of the abdomen and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the antimicrobial properties of one finished test product (ZP) with a positive control (CP) and a negative control (ZP™ Vehicle without IPA) when used as a patient preoperative skin preparation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good health
* Minimum skin flora baseline requirements on abdomen and groin
* Skin free of tattoos, dermatoses, abrasions, cuts, lesions, or other skin disorder near or on the applicable test area.

Exclusion Criteria:

* Topical or systemic antimicrobial exposure within 14 days prior to screening and treatment days, including antibiotics.
* Subjects with a history of skin sensitivity, skin allergies, or skin cancer.
* Subjects who are pregnant, attempting pregnancy or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2017-04-09 (Actual); Study Completion 2017-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, Principal Investigator — Microbac Laboratories, Inc.
Locations (1):
- MicroBioTest Laboratories, Sterling, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edmiston CE, Lavin P, Spencer M, Borlaug G, Seabrook GR, Leaper D. Antiseptic efficacy of an innovative perioperative surgical skin preparation: A confirmatory FDA phase 3 analysis. Infect Control Hosp Epidemiol. 2020 Jun;41(6):653-659. doi: 10.1017/ice.2020.27. PMID 32131912

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment consists of subjects that advanced from screening to randomization and treatment. Each subject had 2 test products applied bilaterally; therefore, the numbers will not add up uniformly across arms due to the pre-determined cohort/block design. Result totals will be less than than the treated number as the per subject/area/intervention anatomical site must have an acceptable baseline count/flora.
Units Other Than Participants: Ab or groin
Groups:
- All Participants: ZP (Isopropyl alcohol (IPA) 70%) or CP or ZP Vehicle Applied topically to ab (for 30 seconds) or groin (for 2 minutes).
Period: Overall Study
Arm/Group | All Participants
Started | 440; 440 Ab or groin
ZP | 400; 400 Ab or groin
CP | 400; 400 Ab or groin
Vehicle | 80; 80 Ab or groin
Completed | 440; 440 Ab or groin
Not Completed | 0; 0 Ab or groin

BASELINE CHARACTERISTICS:
Groups:
- Treated Population: Each subject could have received 2 out of 3 test products randomly assigned. Demographics were not stratified by test product due to study design. While 440 was the treated population, to be evaluable for efficacy, each subject anatomical sample site (4/per subject) would need to pass the minimum log10 baseline requirements.
Arm/Group | Treated Population
Number analyzed (Participants) | 440
Age, Continuous [Mean (Full Range); unit: years] | 38.4 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45
  Not Hispanic or Latino | 379
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 119
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 84
  White | 176
  More than one race | 0
  Unknown or Not Reported | 61

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Reduction
Description: A 3-log10 CFU/cm^2 bacterial reduction on the inguinal region is considered a success.
Time Frame: 10 minutes post product application
Population: Treated subjects with a treatment day baseline criteria of 5.0-7.5 log10 CFU/cm^2 recoveries for each sampling site (2 groin sampling sites per subject).
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Groups:
- Mean Log Reduction - ZP (70% IPA) - Groin: Isopropyl alcohol (IPA) 70%
  ZP: Apply topically.
- Mean Log Reduction - ChloraPrep - Groin: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically.
- Mean Log Reduction - ZP Vehicle - Groin: ZP without IPA
  ZP Vehicle: Apply topically.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Groin | Mean Log Reduction - ChloraPrep - Groin | Mean Log Reduction - ZP Vehicle - Groin
Number analyzed (Participants) | 330 | 326 | 68
log10 CFU/cm^2 | 4.83 (0.1) | 4.78 (0.1) | 2.23 (0.2)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - ChloraPrep - Groin; Groin 10 minutes Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and the predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product upper bounds must be less than 0.5; Median Difference (Final Values) = -0,052, 95% CI 2-sided [-0.188 to 0.083]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - ZP Vehicle - Groin; Groin 10 minutes Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Superiority — Investigational product lower bounds must be greater than 1.2; Median Difference (Final Values) = 2.627, 95% CI 2-sided [2.396 to 2.858]

2. Primary Outcome: Bacterial Reduction - Abdomen
Description: A 2-log10 CFU/cm^2 bacterial reduction on the abdomen region is considered a success.
Time Frame: 10 minutes post product application
Population: Treated subjects with a treatment day baseline criteria of 3.0 - 5.5 Log10 CFU/cm^2 recoveries.
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Groups:
- Mean Log Reduction - ZP (70% IPA) - Abdomen: Isopropyl alcohol (IPA) 70%
  ZP: Apply topically.
- Mean Log Reduction - ChloraPrep - Abdomen: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically.
- Mean Log Reduction - ZP Vehicle - Abdomen: ZP without IPA
  ZP Vehicle: Apply topically.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Abdomen | Mean Log Reduction - ChloraPrep - Abdomen | Mean Log Reduction - ZP Vehicle - Abdomen
Number analyzed (Participants) | 342 | 340 | 69
Log10 CFU/cm^2 | 3.35 (0.1) | 3.34 (0.1) | 1.47 (0.2)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - ChloraPrep - Abdomen; Abdomen 10 minutes Average Treatment Effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 CFU/cm^2 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 CFU/cm^2 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product average treatment effect upper bounds cannot be more than 0.5; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.102 to 0.065]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - ZP Vehicle - Abdomen; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Investigational product lower bounds must be greater than 1.2; Mean Difference (Final Values) = 1.909, 95% CI 2-sided [1.766 to 2.053]

ADVERSE EVENTS:
Time Frame: 6 hours post product application
Groups:
- ZP (70% IPA): Isopropyl alcohol (IPA) 70%
  ZP: Apply topically.
Arm/Group | ZP (70% IPA) | ChloraPrep | ZP Vehicle
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/400 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/80
Other Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02831998/Prot_SAP_000.pdf